CLINICAL TRIAL: NCT02611154
Title: Intranasal Delivery of Testosterone and Its Effect on Doping Markers
Acronym: Intranasal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Sports Medicine Research and Testing Laboratory (Industry); Partnership for Clean Competition (Other)
Responsible Party: Principal Investigator, Stuart Willick, M.D., University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 84225
Record Dates: First submitted 2015-11-11; First posted 2015-11-20 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Abuse of Anabolic Steroids
Keywords: Healthy Volunteers; Sports Medicine; Men's Health; Athletes; Anti-Doping
MeSH Terms: interventions — Testosterone; Natesto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intranasal Testosterone (Experimental): All participants will be receiving intranasal testosterone and will follow the same study procedures.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Participants will self-administer 11 mg 3x daily, for 5 consecutive days for 4 weeks.
  Other Names: Natesto

SUMMARY:
Hypothesis: Intranasal administration of exogenous testosterone results in a characteristic profile during anti-doping testing, which is different than the profile seen when testosterone is administered into muscle, on skin or under the tongue.

Objective: The investigators aim to characterize the unique steroid doping profile following administration of intranasal testosterone to healthy, active volunteer subjects.

DETAILED DESCRIPTION:
Testosterone is a substance commonly abused in the sporting world despite being banned by all American sports leagues, international federations, and the World Anti-Doping Agency. Current methods employed to detect exogenously administered testosterone include direct detection using isotope ratio mass spectrometry (IRMS) and indirect detection using the athlete biological passport (ABP). However, different formulations of testosterone (oral, transdermal, sublingual, etc) are expected to result in characteristic IRMS profiles, affect the ABP readings in unique ways, and differ in their windows of detection. In 2014, a new formulation of testosterone, Natesto, which is administered intranasally, was FDA approved. Though only approved for medical use, it is expected athletes may use this product, and its effect on steroid doping markers has yet to be determined. Characterization of this detection profile is necessary for confirmation of the exact product being administered in an anti-doping setting. In this study, the investigators aim to understand the effects on the steroid doping profile following a single administration of Natesto to healthy, active volunteers. Windows of detection will be determined for the standard dosing of Natesto, and the effects on ABP markers and IRMS profiles will also be established.

ELIGIBILITY:
Inclusion Criteria:

1. Males between the ages of 18 and 35 years-old who participate in regular, moderate to high intensity physical activity will be recruited for the study.

Exclusion Criteria:

1. Individuals below the age of 18 or greater than the age of 35 on the day of enrollment
2. Individuals who are in a Registered Testing Pool for anti-doping purposes, or individuals who for any reason could be subject to doping control testing.
3. Unwilling to provide blood or urine samples
4. Not actively exercising
5. Individuals with any history of cancer, cardiovascular disease, endocrine abnormalities, renal disease, hepatic disease, neurologic disease or any psychiatric history
6. Individuals with a history of nasal disorders, nasal surgeries, sinus surgeries, or sinus disease
7. Individuals that have a baseline hematocrit value above the normal range
8. Individuals that are diabetic or are currently taking a diabetic medication
9. Individuals that are currently using any WADA prohibited substances
10. Individuals that have recently used or currently using anabolic androgenic steroids

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2016-01-19 (Actual); Study Completion 2016-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Willick, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Data will be published in scientific literature without Patient Health Information (PHI) identifying any participant data.

REFERENCES:
- [Background] Saudan C, Baume N, Robinson N, Avois L, Mangin P, Saugy M. Testosterone and doping control. Br J Sports Med. 2006 Jul;40 Suppl 1(Suppl 1):i21-4. doi: 10.1136/bjsm.2006.027482. PMID 16799097
- [Background] Geyer H, Schanzer W, Thevis M. Anabolic agents: recent strategies for their detection and protection from inadvertent doping. Br J Sports Med. 2014 May;48(10):820-6. doi: 10.1136/bjsports-2014-093526. Epub 2014 Mar 14. PMID 24632537
- [Background] Sottas PE, Saugy M, Saudan C. Endogenous steroid profiling in the athlete biological passport. Endocrinol Metab Clin North Am. 2010 Mar;39(1):59-73, viii-ix. doi: 10.1016/j.ecl.2009.11.003. PMID 20122450
- [Background] Vernec AR. The Athlete Biological Passport: an integral element of innovative strategies in antidoping. Br J Sports Med. 2014 May;48(10):817-9. doi: 10.1136/bjsports-2014-093560. Epub 2014 Mar 21. PMID 24659508
- [Background] Jia H, Sullivan CT, McCoy SC, Yarrow JF, Morrow M, Borst SE. Review of health risks of low testosterone and testosterone administration. World J Clin Cases. 2015 Apr 16;3(4):338-44. doi: 10.12998/wjcc.v3.i4.338. PMID 25879005
- [Background] Bassil N, Alkaade S, Morley JE. The benefits and risks of testosterone replacement therapy: a review. Ther Clin Risk Manag. 2009 Jun;5(3):427-48. doi: 10.2147/tcrm.s3025. Epub 2009 Jun 22. PMID 19707253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study began in November 2015 and ended December 2015. The final participant was enrolled on 03DEC2015 and completed the study on 19JAN2016.
Period: Overall Study
Arm/Group | Intranasal Testosterone
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intranasal Testosterone
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex/Gender, Customized [Number; unit: participants]
  Male Participants | 5
Region of Enrollment [Number; unit: participants] — Salt Lake City, Utah, USA
  participants
    United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Steroid Levels in Urine Steroid Profile
Description: Participants were instructed to follow this dosing pattern:
  Begin taking Intranasal Testosterone at Day 1 for 5 consecutive days (Days 1-5), then to take 2 days off (Day 6 and 7) Urine sample at Day 6 Begin taking Intranasal Testosterone at Day 8 for 5 consecutive days (Days 8-12), then to take 3 days off (Day 13, Day 14, Day 15) Urine sample at Day 13 Begin taking Intranasal Testosterone at Day 16 for 5 consecutive days (Days 16-20), then to take 2 days off (Day 21 and 22) Urine sample at Day 21 Begin taking Intranasal Testosterone at Day 23 for 5 consecutive days (Days 23-27 ), then to take 2 days off (Day 28 and 29) Urine sample at Day 28
  The first day of the dosing pattern is considered Day 1 and the last day of the pattern is considered Day 29.
  Samples 4-8 were analyzed between 0 and 24hours post-dose Sample 9 was analyzed 48 hours post-dose Sample 10 was analyzed 72 hours post-dose Sample 11 was analyzed one week post-dose
Time Frame: 4 weeks of dosing for each participant
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Urine Steroid Profile - Day 6: Day 6 steroid level in urine. Urine sample analyzed within 24 hours of dosing.
- Urine Steroid Profile - Day 13: Day 13 steroid level in urine. Urine sample analyzed within 24 hours of dosing.
- Urine Steroid Profile - Day 21: Day 21 steroid level in urine. Urine sample analyzed within 24 hours of dosing.
- Urine Steroid Profile - Day 28: Day 28 steroid level in urine. Urine sample analyzed within 24 hours of dosing.
- Urine Steroid Profile - Day 29: Day 29 steroid level in urine. Urine sample analyzed within the 24-48 hour window post-administration.
- Urine Steroid Profile - Day 30: Day 30 steroid level in urine. Urine sample analyzed within the 48-72 hour window post-administration.
- Urine Steroid Profile - Day 35: Urine was collected at Day 35 to identify any suppression of endogenous testosterone production following administration.
- Urine Steroid Profile - Day 42: Urine was collected at Day 42 to identify any suppression of endogenous testosterone production following administration.
Arm/Group | Urine Steroid Profile - Day 6 | Urine Steroid Profile - Day 13 | Urine Steroid Profile - Day 21 | Urine Steroid Profile - Day 28 | Urine Steroid Profile - Day 29 | Urine Steroid Profile - Day 30 | Urine Steroid Profile - Day 35 | Urine Steroid Profile - Day 42
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5
ng/mL
  Testosterone | 69.5773456 (35.54601116) | 138.0291641 (141.9066157) | 163.117081 (109.276721) | 107.7160658 (113.703136) | 14.15587072 (4.228012086) | 21.42280994 (14.29364856) | 32.9077285 (13.76180063) | 28.14492389 (6.661553442)
  Epitestosterone | 14.54132527 (7.954646945) | 16.23444899 (11.98868156) | 10.08654906 (4.588211806) | 9.736167767 (4.015340993) | 12.22899541 (4.434891082) | 16.38534782 (4.918171284) | 27.76476978 (16.66310752) | 32.56796986 (10.94213563)
  Androsterone | 2780.422993 (1545.144279) | 3147.357191 (2520.278196) | 3377.718911 (1511.306185) | 4014.439418 (4846.667258) | 1098.544542 (430.6835869) | 1689.228939 (968.2213645) | 2292.971167 (853.7596469) | 1561.824479 (663.1827091)
  Etiocholanolone | 3420.811467 (2957.358109) | 2984.088377 (2078.022714) | 3168.249168 (1630.873996) | 4614.568182 (7192.193898) | 1154.779419 (460.2075499) | 1810.282342 (1552.137347) | 2612.685992 (2105.416619) | 1281.752255 (372.3518874)
  5αAdiol | 81.50246345 (28.87216828) | 70.09892435 (31.91867777) | 79.92660959 (19.82671546) | 83.39693284 (59.00306611) | 37.53345262 (7.673138406) | 51.7003489 (22.77519196) | 60.19484767 (21.91151504) | 56.94343765 (30.25653073)
  5βAdiol | 323.5235566 (95.27658018) | 370.2752839 (244.8399242) | 386.6496467 (178.3061711) | 369.209311 (243.4060107) | 145.5896139 (54.18663296) | 158.5303528 (90.57253904) | 166.0185686 (97.42880397) | 85.54384971 (17.46215146)

2. Secondary Outcome: Number of Participants With Suspicious Steroid Profile in Urine Samples at Baseline
Description: Participants were asked to provide 3 urine samples at Day 1, Day 3, Day 5 to measure their baseline urinary steroid marker levels. To accommodate participant schedules, all baseline samples were collected within a two week timeframe. This outcome is measuring if any participants baseline urine samples resulted in a suspicious steroid profile. For this study, "suspicious" is defined as any urine sample resulting in testosterone steroid detection above 200ng/mL.
Time Frame: Day 1, Day 3, Day 5
Measure: Count of Participants; unit: Participants
Groups:
- Testosterone: Testosterone level will be measured in the urine sample.
- Epitestosterone: Epitestosterone level will be measured in the urine sample.
- Androsterone: Androsterone level will be measured in the urine sample.
- Etiocholanolone: Etiocholanolone level will be measured in the urine sample.
- 5αAdiol: 5αAdiol level will be measured in the urine sample.
- 5βAdiol: 5βAdiol level will be measured in the urine sample.
Arm/Group | Testosterone | Epitestosterone | Androsterone | Etiocholanolone | 5αAdiol | 5βAdiol
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Testosterone Level in Blood as Measured for Safety
Description: Testosterone level in blood to ensure safety levels of testosterone prior to (Day 0) and after the first two weeks of drug administration (Day 19). Steroid levels below the normal range were considered safe to continue study participation.
Time Frame: Day 0 and Day 19
Measure: Mean (Full Range); unit: ng/mL
Groups:
- Serum Testosterone - Day 0: Serum Testosterone at Day 0
- Serum Testosterone - Day 19: Serum Testosterone at Day 19
Arm/Group | Serum Testosterone - Day 0 | Serum Testosterone - Day 19
Number analyzed (Participants) | 5 | 5
ng/mL | 408.4 [300 to 1080] | 373.4 [300 to 1080]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Intranasal Testosterone
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No